CLINICAL TRIAL: NCT01302769
Title: Ear Acupuncture for Acute Sore Throat. A Randomized Controlled Trial.
Brief Title: Ear Acupuncture for Acute Sore Throat.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWH20110008H
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Acute Sore Throat
Keywords: Acute Sore Throat; Ear Acupuncture
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- battlefield auricular acupuncture (Experimental): battlefield auricular acupuncture
  Interventions: Device: Standard treatment plus ear acupuncture
- placebo (No Intervention)

INTERVENTIONS:
Device: Standard treatment plus ear acupuncture — Standard treatment plus ear acupuncture
  Other Names: Sedatelec ASP Original Gold needles
  Arms: battlefield auricular acupuncture

SUMMARY:
The purpose of this study is to compare ear acupuncture plus standard of care versus standard therapy (anti-inflammatory medications) in the reduction of pain, reduction in oral anti inflammatory medication use, hours lost from work in acute sore throat.

ELIGIBILITY:
Inclusion:

* Male and female subjects (DoD beneficiaries), 18 years or older, with upper respiratory complaints and their primary symptom being acute sore throat.
* Minimum pain score of 5 points on an 11 point scale (0-10 with 10 being the worst pain)

Exclusion:

* History of significant gastrointestinal bleed
* Previous documented history of stage 2 kidney disease or worse
* Known Pregnancy
* History of gastric bypass surgery
* Known Peritonsillar abscess (PTA)
* Throat, mouth or esophageal cancer
* Chronic oral steroids use
* Absence of one or more ears
* Active cellulitis of ear
* Ear anatomy precluding identification of acupuncture landmarks
* Non-English speaking
* Use of Hearing Aids that preclude the use of ear acupuncture
* Allergy to Ibuprofen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Moss, M.D., Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (1):
- Mike O'Callaghan Federal Hosptial, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Not permitted to share data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: standard of care
Period: Overall Study
Arm/Group | Battlefield Auricular Acupuncture | Placebo
Started | 28 | 28
Completed | 27 (analyzed) | 27 (analyzed)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: 28 were initially in study. Each arm lost one subject to follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Battlefield Auricular Acupuncture | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Control- 1 patient lost to follow up Intervention- 1 patient lost to follow up
  Participants
    Female | 15 | 20 | 35
    Male | 12 | 7 | 19
throat culture [Count of Participants; unit: Participants] — If throat culture is positive, patients will be notified and referred to their Primary Care Manager to be prescribed standard of care antibiotics
  Participants | 0 | 0 | 0
urine pregnancy test [Count of Participants; unit: Participants] — If there is a chance that the subject could be pregnant, they will be sent for a urine pregnancy test (15-20 mls or approximately 2-3 teaspoons of urine).
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Pain
Description: Subjects will be randomized to receive either standard treatment alone or standard treatment plus ear acupuncture.
  Subjects will be asked 15 minutes after their treatment to assess their pain on a likert scale of 0-10. After the subject has left the clinic, phone calls will be made at 6 hours, 24 hours and 48 hours to assess their pain level.
  Scale: 11-point scale of 0-10 with 10 being the worst pain.
  Subjects who report back after 48 hours with unimproved sore throat will be instructed to make a same day follow up with the clinic.
Time Frame: 48 hours per subject
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Battlefield Auricular Acupuncture | Placebo
Number analyzed (Participants) | 27 | 27
score on a scale
  Pain scores (0-10) [0 minutes] | 6.4 [6.0 to 6.8] | 6.2 [5.7 to 6.7]
  Pain scores (0-10) [15 minutes] | 2.6 [1.7 to 3.5] | 6.0 [5.4 to 6.6]
  Pain scores (0-10) [6 hours] | 2.5 [1.6 to 3.4] | 4.8 [4.0 to 5.6]
  Pain scores (0-10) [24 hours]] | 1.9 [1.0 to 2.8] | 4.1 [3.3 to 4.9]
  Pain scores (0-10) [48 hours]] | 1.3 [0.6 to 2.0] | 2.3 [1.6 to 3.0]

2. Primary Outcome: Ibuprofen Doses Taken
Description: Subjects will be randomized to receive either standard treatment alone or standard treatment plus ear acupuncture.
  After the subject has left the clinic, phone calls will be made at 6 hours, 24 hours and 48 hours to ask the number of doses of ibuprofen taken.
Time Frame: 48 hours per subject
Measure: Mean (95% Confidence Interval); unit: number ibuprofen doses taken
Arm/Group | Battlefield Auricular Acupuncture | Placebo
Number analyzed (Participants) | 27 | 27
number ibuprofen doses taken
  ibuprofen doses taken (6 hours) | 0.39 [0.2 to 0.58] | 1.07 [0.69 to 1.45]
  ibuprofen doses taken (24 hours) | 1.37 [0.92 to 1.82] | 2.63 [1.95 to 3.31]
  ibuprofen doses taken (48 hours) | 2.19 [1.44 to 2.94] | 4.07 [2.9 to 5.24]

3. Primary Outcome: Missed Work Hours
Time Frame: 48 hours per subject
Measure: Mean (95% Confidence Interval); unit: number hours missed from work
Arm/Group | Battlefield Auricular Acupuncture | Placebo
Number analyzed (Participants) | 27 | 27
number hours missed from work
  Missed work hours [15 minutes] | 0.61 [0.0 to 1.25] | 1.13 [0.49 to 1.77]
  Missed work hours [6 hours] | 1.57 [0.66 to 2.48] | 3.19 [1.91 to 4.47]
  Missed work hours [24 hours] | 3.04 [1.34 to 4.74] | 5.48 [3.25 to 7.71]
  Missed work hours [48 hours] | 3.78 [1.63 to 5.93] | 6.48 [3.99 to 8.97]

ADVERSE EVENTS:
Time Frame: 48 hours (per subject)
Description: No difference.
Arm/Group | Battlefield Auricular Acupuncture | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

LIMITATIONS AND CAVEATS:
Small sample size, no sham acupuncture, subjects not blinded to treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study takes place at military hospital with DoD active duty, veterans, and beneficiaries. Publishing of aggregate or simply deidentified data is prohibited.